CLINICAL TRIAL: NCT06274476
Title: Short-Term Evaluation of Prosthetic Rehabilitation of Thin Wiry Ridge by Ridge Splitting and Simultaneous Implants Placement: Non-randomized Control Trial
Brief Title: Prosthetic Rehabilitation of Thin Wiry Ridge by Ridge Splitting and Simultaneous Implants Placement
Acronym: implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020/9/9
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Atrophic Maxillary Ridge and Mandibular Ridge
Keywords: implant; knife-edge ridge; ridge expansion; piezoelectric; implant-supported prosthesis; prosthetic complications

STUDY DESIGN:
Intervention Model Description: maxillary and mandibular atrophic ridge
Who Masked: Investigator, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxillary atrophic ridge (Experimental): received ridge splitting done by piezo surgery and implant placement in maxillary arch
  Interventions: Other: implant placement
- mandibular atrophic ridge (Active Comparator): received ridge splitting done by saw technique using ridge expanders and implant placement in maxillary arch
  Interventions: Other: implant placement

INTERVENTIONS:
Other: implant placement — ridge splitting piezo surgery and implant placement
  Other Names: implant installation

SUMMARY:
evaluates the success of prosthetic rehabilitation of thin wiry ridge and implants placed simultaneously in splitted ridge both clinically and radiographically.

DETAILED DESCRIPTION:
twenty-one participants were enrolled of which 13 patients (8 females and 5 males) were suffering from maxillary ridge atrophy and 8 patients (5 females and 3 males) had mandibular ridge atrophy; a total of 42 implants were performed using the ridge expansion technique. The expansion was performed using the conventional disk technique, piezoelectric corticotomy, and self-threading expanders. Implants were placed and loaded with fixed partial denture after 4 months for the mandible and 6 months for the maxilla. Implant stability quotient (ISQ) was measured at T0 (implant placement) and TL (loading). Crestal bone levels were measured at different times: T0, TL, and T12 (12 months). Evaluation of prosthetic and surgical complications was carried out. Data were analyzed and compared using analysis of variance and paired t-tests at a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* ridge of 2 to 4 mm of initial alveolar crest width
* bone height of at least 8 mm from vitastructures

good oral hygiene.

Exclusion Criteria:

patients who smoke more than 10 cigarettes per day diabetes mellitus, osteoporosis, and periodontal disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
implant success | 12 month
  implant osseointgeration by radiographic evaluation .bone loss by mm, and bone density

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed yahia Sharaf, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No